CLINICAL TRIAL: NCT03478579
Title: Nontechnical Skills Assessment of Emergency Physicians and Quality of Care in a Virtual Emergency Department
Brief Title: Non-technical Skills of Emergency Physicians in a Virtual Emergency Department
Acronym: 3D-QUAMU
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC 31/16/8763
Record Dates: First submitted 2017-06-08; First posted 2018-03-27 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Emergencies
Keywords: serious game; simulation; virtual emergency department; nontechnical skills
MeSH Terms: conditions — Emergencies | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Emergency physicians: The observational group will be composed of emergency physicians working in the French Midi-Pyrenees region. Physicians must work since 2 years in emergency service
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — No intervention, it is observational study

SUMMARY:
The investigators will study nontechnical skills of emergency physicians in a virtual standardized emergency room and their impact on quality of care.

DETAILED DESCRIPTION:
The ability to manage multiple patients and anticipate the risk of error related to task interruptions or disruptions has been identified among relevant non-technical skills (NTS) for practicing emergency medicine. However, the link between these skills and the quality of care has not been quantified. NTS are usually analyzed by qualitative methods such as interviews, direct observations, or questionnaires that have low performance according to the GRADE system (Grading of Recommendations, Assessment, Development and Evaluation).

The investigators have created and validated an experimental model of a virtual, authentic and realistic Emergency Department (ED). The platform has been modelled in a "Second Life" environment. The NTS of emergency physicians will be assessed and recorded during simulated care of multiple virtual patients. The NTS association with ED length of stay and disposition decision will be analyzed. This study will be an internal pilot study and will include 30 emergency physicians who practice emergency medicine for at least two years.

Sessions will be performed in the Toulouse Institute of Health Care Simulation, Toulouse University Hospital. They will be composed of three stages: briefing (30 minutes), simulated practice (3 hours), and debriefing with an explicit interview (30 minutes). Two researchers and a computer technician will supervise the sessions. The data will be obtained by analyzing the video recorded during the simulated practice and the interview.

ELIGIBILITY:
Inclusion Criteria:

* Active emergency physicians working in an ED of the French Midi-Pyrenees region
* Two years of practice in emergency medicine or more
* Volunteer to participate in the study

Exclusion Criteria:

* Emergency physician working in another setting than ED, outside the Midi-Pyrenees region, or practicing emergency medicine for less than 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Emergency physicians working in the French Midi-Pyrénées region
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Nontechnical skills | 3 hours
  The nontechnical skills will be assessed by the Anaesthetists' Non-Technical Skills (ANTS) system.

SECONDARY OUTCOMES:
Quality of care will be measured by a composite criteria (process and result) | 3 hours
  Quality of care will be measured by a composite criterion associating a process indicator and a result indicator :
  * The process indicator is the average time to medical care of patients
  * The result indicator corresponds to the relevance of the choice of the orientation of each patient by the emergency doctor at the end of medical care
ED length of stay | 3 hours
  The quality of care will be assessed by ED length of stay : ED length of stay will be measured from triage completion to disposition decision
The authenticity of the virtual emergency medicine service | 3 hours
  Evaluation of the consistency : perceived internal consistency in the proposed rules and situations will be assessed using a 4-item questionnaire by answering yes or no
The authenticity of the virtual emergency medicine service | 3 hours
  Evaluation of the realism (the assumed resemblance with a real life reference) will be evaluated through a questionnaire containing 3 areas of comparison between the virtual and real environment (layout of the premises, duration of the actions, staff / patient ratio) with as answer possible for each comparison: Realistic or not realistic.
The authenticity of the virtual emergency medicine service | 3 hours
  Evaluation of the relevance (necessary to allow users to take ownership of the problems posed by the designers) will be assessed through direct observation with a yes / no evaluation of the acceptance to use the virtual environment, to test the environment, to make choices during the scenario and to control the environment.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Lauque, MD, Study Chair — Toulouse CHU
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No